CLINICAL TRIAL: NCT03118115
Title: Bioimpedance Variation of Free Flap for After Clamping - MONITRANS
Brief Title: Bioimpedance Variation of Free Flap for After Clamping
Acronym: MONITRANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2016_843_0028
Record Dates: First submitted 2017-03-22; First posted 2017-04-18 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Thrombosis
Keywords: bioimpedance; thrombosis; free flap; microsurgerie; breast reconstruction
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Intervention Model Description: Measurement of the flap bioimpedance before and after clamping of the artery or the vein. For information: All patients will have the vein and the arterial section simulating venous or arterial thrombosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impedance (Experimental): Measurement of the flap bioimpedance before and after clamping of the artery or the vein. For information: All patients will have the vein and the arterial section simulating venous or arterial thrombosis.
  Interventions: Device: Measurement of the flap bioimpedance

INTERVENTIONS:
Device: Measurement of the flap bioimpedance — Measurement of the flap bioimpedance before and after clamping of the artery or the vein. For information: All patients will have the vein and the arterial section simulating venous or arterial thrombosis.

SUMMARY:
MONITRANS project consist of developing a monitoring technology of post-operative breast reconstruction by detecting thrombosis. Its aim is to reducing time spent in hospital by monitoring patients at home.

Thrombosis following to abdominal free flap harvesting for breast reconstruction is a rare phenomenon (with a 2 until 15 % frequency). Moreover, it leads to ischemia by limiting water intake in the plasma compartments. The investigator would like to prove, by this research project, that they are able to detect ischemia via bioimpedance technology.

During abdominal free flap harvesting for breast reconstruction, there are few minutes where the flap is clamped because of anastomosis on the recipient vessels. The investigators would seize the opportunity of this step, which is similar to vascular thrombosis, to measure bioimpedance variations.

Therefore they would like to measure variations of the flap bioimpedance before and after vascular section. Another purpose consists of developing an algorithm which will detect postoperative thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* patient suitable for a abdominal perforator based flap breast reconstruction
* age over 18 years old

Exclusion Criteria:

* pregnancy
* women with active pacemaker implant or artificial heart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Measurement of impedence | 1 day
  Measurement of the flap bioimpedance before and after clamping of the artery or the vein.

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël SINNA, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No